CLINICAL TRIAL: NCT06136104
Title: The Effects of Mixhers HERTIME Supplements on Menstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 23007
Record Dates: First submitted 2023-10-27; First posted 2023-11-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Premenstrual Dysphoric Disorder; Premenstrual Syndrome
Keywords: PMS (Premenstrual syndrome); PMDD (Premenstrual dysphoric disorder); Period Symptoms; Menstrual Cycle; Menstrual Cramping; Menstrual Bleeding
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixhers HERTIME (Experimental): 1 daily powder stick packet (3.0-3.3 g) of Mixhers HERTIME herbal supplement mixed into water
  Interventions: Dietary Supplement: Mixhers HERTIME
- Placebo (Placebo Comparator): 1 daily powder stick packet (3 g) of a matching placebo powder supplement mixed into water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mixhers HERTIME — A daily self-administered powder supplement packet mixed into water.
  Arms: Mixhers HERTIME
Dietary Supplement: Placebo — A daily self-administered powder placebo supplement packet mixed into water.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess Mixhers HERTIME supplements efficacy in alleviating menstrual cycle symptoms.

DETAILED DESCRIPTION:
All participants, after providing written informed consent, will drink a daily self-administered powder-mix supplement in water of either placebo or Mixhers HERTIME for 120 consecutive days. Surveys will be administered electronically to each participant in the first month to assess baseline menstrual cycle symptoms. In addition, before starting the supplement, participants will take the electronic survey "The Premenstrual Symptoms Screening Tool". During the first month of taking the supplement, participants will take an allergy and constitutional symptom survey electronically to assess for any adverse reactions to the product. Each month for four months, participants will complete an electronic survey assessing menstrual cycle symptoms after a menstrual cycle is completed.

ELIGIBILITY:
Inclusion Criteria:

* Must be biologically female, must have a regular menstrual cycle (defined as a menstrual bleed every 23-35 days), must be a student, staff, or faculty member at Midwestern University Glendale, Arizona campus

Exclusion Criteria:

* not pregnant or planning to become pregnant, must not be on anticoagulants, must not have allergies to lemon or stevia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Menstrual Cramping and/or Back Pain | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Mood Regulation | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 mood scale
Bloating | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Menstrual Bleeding Volume | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 scale of flow volume
Menstrual Bleeding Duration | 120 days
  Measured through post-menstrual bleeding electronic survey recording start and end day of menstrual bleeding

SECONDARY OUTCOMES:
Fatigue | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 scale of fatigue experienced
Acne | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Difficulty Concentrating | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Overeating/Food Cravings | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Insomnia | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Hypersomnia | 120 days
  Measured through post-menstrual bleeding electronic survey 1-10 severity scale
Period symptom interference with school/work efficiency/productivity | 120 days
  Measured through post-menstrual bleeding electronic survey four-point Likert scale
Period symptom interference with social life activities | 120 days
  Measured through post-menstrual bleeding electronic survey four-point Likert scale
Period symptom interference with physical activity (sports, gym, or daily performance) | 120 days
  Measured through post-menstrual bleeding electronic survey four-point Likert scale
Any positive or negative mood changes noticed during period | 120 days
  Measured through post-menstrual bleeding electronic survey free response prompt
Any positive or negative mood changes noticed during other weeks of the menstrual cycle not bleeding | 120 days
  Measured through post-menstrual bleeding electronic survey free response prompt
Non-steroidal anti-inflammatory drug use for acute symptoms during menstrual bleeding | 120 days
  Measured through post-menstrual bleeding electronic survey free response prompt
Number of pads/tampons/other products used during menstrual bleeding | 120 days
  Measured through post-menstrual bleeding electronic survey free response prompt

OTHER OUTCOMES:
Other miscellaneous changes noticed during menstrual bleeding | 120 days
  Measured through post-menstrual bleeding electronic survey free response prompt

CONTACTS AND LOCATIONS:
Overall Officials: Farshad Agahi, MD, Principal Investigator — Midwestern University- Glendale, AZ
Locations (1):
- Midwestern University, Glendale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No